CLINICAL TRIAL: NCT00370916
Title: Reducing Transition Drug Risks After Patient Transfer
Brief Title: Reducing Transition Drug Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Victoria (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IAB 05-204
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2010-12

CONDITIONS: Hospitalization
Keywords: Clinical Decision Support Systems; Continuity of Patient Care; Medication Errors; Drug Adverse Effects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Physician-initiated medication reconciliation
  Interventions: Behavioral: Physician-initiated medication reconciliation
- Arm 2 (Experimental): Pharmacist-initiated medication reconciliation
  Interventions: Behavioral: Pharmacist-initiated medication reconciliation
- Arm 3 (No Intervention): No formal medication reconciliation

INTERVENTIONS:
Behavioral: Physician-initiated medication reconciliation — Physician house staff performed and documented medication reconciliation after hospital admission with the assistance of a CPRS template
  Arms: Arm 1
Behavioral: Pharmacist-initiated medication reconciliation — Pharmacist performed and documented medication reconciliation
  Arms: Arm 2

SUMMARY:
Patient transfer between sites of care is regular practice during an episode of care in our current health care system. Yet inter-site transfer is associated with lapses in care quality that adversely affect patient outcomes. A common iatrogenic harm precipitated at the time of transfer is harm from drug prescribing, or adverse drug events (ADEs). In this study we will evaluate a medication reconciliation tool developed to help providers make effective prescribing decisions at the time of transfer between VA sites of care (Improved Prescribing after Transfer (IPT)). We will evaluate the quantitative effectiveness of the tool in reducing transition drug risk and ADEs. We additionally will conduct focus group discussions and cognitive task analysis among end-users to better understand how providers make drug-prescribing decisions at the time of transfer and to assess factors influencing effective use of the tool.

DETAILED DESCRIPTION:
This is a 2-phase study in which we will employ mixed quantitative and qualitative methods to conduct an evaluation of the IPT tool while improving our understanding of provider prescribing decisions at the time of patient transfer. In Phase 1 we will conduct a 5-month controlled trial among all admissions to 2 units at J.J. Peters (Bronx) VA Medical Center. We will compare IPT with usual care, and compare physician and pharmacist forms of IPT implementation with regard to, as primary outcome, transition drug risk, and, as secondary outcomes, ADEs, provider prescribing-decisions, and hospital utilization. In Phase 2, which will run concurrently with Phase 1, we will perform cognitive task analysis to examine providers' decision-making and to map IPT tool functions while providers interface with the tool, and perform focus group interviews with representative IPT users to identify factors that facilitate or hinder adoption. Results of cognitive analysis and focus groups will be used to identify tool deficiencies to consider for redesign.

ELIGIBILITY:
Inclusion Criteria:

All patients who were admitted to the JJ Peters (Bronx) VA Hospital general medical wards (units 7A and 7B) between 10/05-2/06 and stayed least 24 hours

Exclusion Criteria:

Patients who were transferred to one of the study units wards (units 7A and 7B) from another JJ Peters (Bronx) VA Hospital acute care unit (e.g., an intensive care unit), or who stayed in the hospital less than 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
High risk drug discrepancies | After hospital admission and discharge

SECONDARY OUTCOMES:
Drug discrepancy adverse events | During the hospital stay and 1 month after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Boockvar, MD MS, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

REFERENCES:
- [Result] Boockvar KS, Santos SL, Kushniruk A, Johnson C, Nebeker JR. Medication reconciliation: barriers and facilitators from the perspectives of resident physicians and pharmacists. J Hosp Med. 2011 Jul-Aug;6(6):329-37. doi: 10.1002/jhm.891. PMID 21834114
- [Result] Kushniruk AW, Santos SL, Pourakis G, Nebeker JR, Boockvar KS. Cognitive analysis of a medication reconciliation tool: applying laboratory and naturalistic approaches to system evaluation. Stud Health Technol Inform. 2011;164:203-7. PMID 21335711
- [Result] Boockvar KS, Blum S, Kugler A, Livote E, Mergenhagen KA, Nebeker JR, Signor D, Sung S, Yeh J. Effect of admission medication reconciliation on adverse drug events from admission medication changes. Arch Intern Med. 2011 May 9;171(9):860-1. doi: 10.1001/archinternmed.2011.163. No abstract available. PMID 21555668
- [Derived] Mergenhagen KA, Blum SS, Kugler A, Livote EE, Nebeker JR, Ott MC, Signor D, Sung S, Yeh J, Boockvar KS. Pharmacist- versus physician-initiated admission medication reconciliation: impact on adverse drug events. Am J Geriatr Pharmacother. 2012 Aug;10(4):242-50. doi: 10.1016/j.amjopharm.2012.06.001. Epub 2012 Jul 20. PMID 22819386